CLINICAL TRIAL: NCT03066544
Title: Status Migrainosus - Differentiating Between Responders and Non-responders in the Setup of Real-life Clinical Practice
Brief Title: Status Migrainosus - Differentiating Between Responders and Non-responders
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hartford HealthCare (Other)
Responsible Party: Principal Investigator, David O'Sullivan, statistician/senior scientist, Hartford HealthCare
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HHC-2016-0221
Record Dates: First submitted 2017-02-21; First posted 2017-02-28 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Migraine
Keywords: migraine; responder; non-responder; treatment
MeSH Terms: conditions — Migraine Disorders | interventions — Bupivacaine; naratriptan; Dexamethasone; Calcium Dobesilate; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Intervention Model Description: This will be a prospective, non-blinded, non-randomized, proof-of-concept study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- bupivacaine (Exparel) (Active Comparator): subjects assigned by clinician's judgment - standard care choice A
  Interventions: Drug: Bupivacaine
- naratriptan pill (Amerge) (Active Comparator): subjects assigned by clinician's judgment - standard care choice B
  Interventions: Drug: Naratriptan Pill
- dexamethasone tablet (Decadron) (Active Comparator): subjects assigned by clinician's judgment - standard care choice C
  Interventions: Drug: Dexamethasone
- ketorolac (Toradol) (Active Comparator): subjects assigned by clinician's judgment - standard care choice D
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Bupivacaine — Nerve blocks with bupivacaine will be performed at initial visit
  Other Names: Exparel
  Arms: bupivacaine (Exparel)
Drug: Naratriptan Pill — one pill will be administered twice each day for 5 days
  Other Names: Amerge
  Arms: naratriptan pill (Amerge)
Drug: Dexamethasone — one tablet will be administered twice each day for 3 days
  Other Names: Decadron
  Arms: dexamethasone tablet (Decadron)
Drug: Ketorolac — ketorolac will be administered intramuscularly (IM) or intravenously (IV) at initial visit
  Other Names: Toradol
  Arms: ketorolac (Toradol)

SUMMARY:
The main goal of this study is to determine whether it is possible - in the setup of routine clinical care - to identify in individual patients who are clear responders to drug X, common denominators that are absent in individual patients who are non-responders to the same drug, and vice versa. All currently available knowledge about migraine pathophysiology will be utilized, using as much time as is needed to ask as many questions as are necessary, in an attempt to profile clear responders and clear non-responders.

DETAILED DESCRIPTION:
Recently, there has been a major focus on "evidence-based" treatments. Who could possibly argue against basing decisions on data? Since the highest level of evidence is derived from randomized double-blind controlled therapeutic trials that consider treatments rendered to large groups of patients with general diagnoses (e.g., migraine) or from a systematic review of several randomized controlled trials (meta analysis), physicians have always prided themselves on applying some type of evidence in order to select treatment. One does not want to imagine medical treatment that is purely subjective. The question, however, is how well does the evidence from trials applies to the care of individual patients? The main problem with such FDA-guided therapeutic trials is the issue of numbers vs specificity. For results to be statistically and biologically valid and important, they must include hundreds and often thousands of participants. To achieve numbers, a lumping strategy predominates over splitting. The more a trial lumps together diverse subgroups, the less specific are the results for individual patients. Given that trials have extensive inclusion and exclusion criteria, often 5 to 10 patients are screened for each patient finally enrolled in the study. Patients who are too ill, too old, too young, female and of childbearing age, incapable of giving informed consent, too complex, or too full of coexisting illnesses are often excluded from trials. Yet, these are the patients who frequently visit the headache center and to whom individualized medicine can provide the most appropriate answers.

Trials that study migraine prevention measure pain intensity and duration, attack frequency, functional disability, quality of life, number of working days lost, nausea, vomiting, and hypersensitivity to light and noise. Whether these measures are those most representative of the important aspects of a condition is an important consideration since not all end points are comparable. Some patients make their living talking. How can their aphasia (difficulty finding the right words) be compared to sensitivity to light or facial numbness? For some patients, it is the sharp pain that continuously pierces through their eyes that makes the headache impossible to tolerate whereas for others it is the ongoing nausea that prevents them from the pleasure of enjoying food, or perhaps the extreme photophobia that makes reading or working on a computer impossible and forces them to quit their jobs and seek the comfort of darkness. How is it, then, that identical weights are assigned to various patients? Physicians are not compelled to treat all patients with a given condition according to identical guidelines, as is the case in therapeutic trials that follow strict protocols. Randomized trials mandate that many patients with a general condition must be given treatment A, and the results are then compared with those of patients given treatment B or C, or placebo. Physicians, however, while caring for one patient at a time must consider several variables, including:

(1) the patient's medical problem; (2) the patient's disease risks; (3) the background, genetics, socioeconomic milieu, psychology, responsibilities, goals, and other characteristics of the patient; and (4) the benefits and risks of potential therapeutic strategies to treat the patient's conditions and to prevent conditions that he or she is at risk of developing.

An inescapable conclusion is therefore that the results of FDA-approved clinical trials fall short of allowing us to 'tailor' the right treatment to the right patient as it does not allow us to predict whether the patient we treat today will or will not benefit from an approved treatment. This conclusion questions the do-ability of translating the often stated goal of individualizing medicine from words to deeds.

Accordingly, the main goal of this proposal is determine whether it is possible - in the setup of routine clinical care - to identify in individual patients who are clear responders to drug X, common denominators that are absent in individual patients who are non-responders to the same drug, and vice versa. All currently available knowledge about migraine pathophysiology will be utilized, using as much time as is needed to ask as many questions as are necessary, in an attempt to profile clear responders and clear non-responders.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* ≥18 years old with no upper age limit
* patients with status migrainosus - defined as a severe migraine headache without aura lasting longer than 72 hours and considered primarily as a complication of migraine
* patients who are willing and able to provide written, informed consent

Exclusion Criteria:

* <18 years old
* unable or unwilling to provide written, informed consent
* females who are pregnant, breastfeeding, or who are trying to become pregnant
* patients who do not speak English
* any medical condition or other reason that in the opinion of the investigators makes the patient unfit or at risk to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11-30 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
time to headache relief | first week
  time to headache relief

CONTACTS AND LOCATIONS:
Overall Officials: Brian Grosberg, MD, Principal Investigator — physician
Locations (1):
- Hartford HealthCare Headache Center, Wethersfield, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No